CLINICAL TRIAL: NCT06497192
Title: Examination of Occupational Justice, Activity Performance and Quality of Life in Homeless People
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Sumeyye Sarısahin, Research Assistant, Bezmialem Vakif University
Other Study IDs: BEZMİALEM-SARIŞAHİN-2024-0001
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Homeless Persons
Keywords: Homelessness; Activitiy performance; Occupational justice; Quality of life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This concerns the participation of individuals experiencing homelessness, as a disadvantaged group, in meaningful and purposeful occupations, evaluated within the framework of occupational justice. Homeless individuals face numerous social and economic barriers that impact their full participation in societal occupations. However, since survival becomes the primary goal for homeless individuals, meaningful occupations often revolve around surviving on the streets. The aim is to identify problems and constraints to participation in daily life activities so that their participation can be enhanced.

DETAILED DESCRIPTION:
"The data collection tools will be implemented during face-to-face interviews with participants. Interview durations will vary between 45 to 90 minutes. Interviews with individuals who accept the invitation to participate will be conducted in public places such as cafes, parks, and other community areas in the Beyoğlu district. The data collection process, initiated after ethical approval, will be concluded upon reaching a sufficient number of participants. Homeless individuals contacted through the 'Çorbada Tuzun Olsun Derneği' will be informed about the research and invited to participate. Individuals with neurological or psychiatric conditions that hinder communication and collaboration will not be included in the study. Fourteen homeless individuals aged 18 or older, literate, able to communicate and collaborate, and currently living on the European side of Istanbul will be included in the study. Data collection instruments for the study include a Demographic Information Form, Semi-Structured Interview Guide, Canadian Occupational Performance Measure, Occupational Justice Health Questionnaire, World Health Organization Quality of Life Scale Short Form, and Occupational Balance Questionnaire."

ELIGIBILITY:
Inclusion Criteria:

* Fourteen homeless individuals aged 18 or older, literate, able to communicate and collaborate, and currently living on the European side of Istanbul will be included in the study.

Exclusion Criteria:

* Individuals with neurological or psychiatric conditions that hinder communication and collaboration will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Homeless individuals
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | Temel
  Measures Demographic Information. It is a form that includes qualitative questions and checklists to assess individuals' current status regarding demographic data such as age, gender, education level, etc.
Semi-Structured Interview Guide | Temel
  Measures living conditions. It includes 4 open-ended questions.
Canadian Occupational Performance Measure | Temel
  Measures Occupational Performance. Self-care, productivity, and leisure constitute three sections. In the initial stage of evaluation, daily life activities identified by the individual are assessed in order of importance on a scale of 1 to 10 (1: not important at all, 10: very important). In the next stage, the individual selects the five most important activities for themselves and is asked to determine performance and satisfaction scores for each activity using a Likert scale from 1 to 10 (1: very poor performance / very dissatisfied, 10: very good performance / very satisfied). The obtained performance and satisfaction scores are summed and divided by the number of activities identified as important by the individual to obtain the performance and satisfaction scores.
Occupational Justice Health Survey | Temel
  Measures Occupational Justice. It is a five-section assessment tool comprising a total of 27 items, addressing fundamental needs, social, physical, and mental well-being, standards of living, and specific injustices that reduce occupational engagement.
World Health Organization Quality of Life Scale Short Form | Temel
  Measures Quality of Life. Since each domain independently represents the quality of life in its own area, domain scores are calculated between 4 and 20. As scores increase, life quality improves.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Sarışahin, MSc, Principal Investigator — Bezmialem Vakıf Üniversitesi
Locations (1):
- Bezmialem Vakıf Üniversitesi, Istanbul, Turkey (Türkiye)